CLINICAL TRIAL: NCT02506478
Title: Journey to Understand and Interpret Juice Preference in the Emergency Department
Brief Title: Juice Preference in the Emergency Department
Acronym: JUICED
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Associate Research Director, Hennepin Healthcare Research Institute
Other Study IDs: 15-3980
Record Dates: First submitted 2015-06-15; First posted 2015-07-23 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: All Eligible ED Patients (Not Limited to a Particular Condition)

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED patients: All ED patients who are able to drink water/juice, and be able to communicate juice preference.
  Interventions: Other: Beverage procurement

INTERVENTIONS:
Other: Beverage procurement — All Emergency Department patients will be approached to ask their beverage preferences in a randomly permuted data collection form. If they would like juice, the flavor will be recorded and the juice (and/or water) will be procured by a research assistant if the patient would like that, though the actual procurement of the juice is not part of the study.

SUMMARY:
ED patients who are able to drink juice will be approached and asked their beverage preference.

DETAILED DESCRIPTION:
Once per week for 26 weeks, patients will be enrolled during a randomly selected 1-hour block. The random blocks will be assigned using STATA. During these enrollment periods, all current ED patients will be screened by the treating physicians and research associates, excluding patients in the "Special Care" unit, where most patients are intoxicated with alcohol.

Eligibility for oral consumption of water and juice will be determined by treating physicians. Patients who are deemed eligible to drink water or juice will be approached and asked their beverage preferences. Their response will be recorded, and the beverage will be procured for them.

ELIGIBILITY:
Inclusion Criteria:

* All Emergency Department patients, of any age, who are cleared by their treating physician to drink juice, and are able to communicate a juice preference. Patients are only enrolled during randomly selected 1-hour blocks once per week for 26 weeks.

Exclusion Criteria:

* Previously enrolled in the study
* Patients who are placed in the "special care" unit of the Emergency Department, which generally cares for intoxicated patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Emergency Department patients, of any age, who are cleared by their treating physician to drink juice, and are able to communicate a juice preference.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Juice preference | 1 hour
  Cranberry, apple, orange, or grape

SECONDARY OUTCOMES:
Beverage preference | 1 hour
  Water, juice, or both
Ice preference | 1 hour
  Yes or no (in any beverage)
Alternate juice preference | 1 hour
  For those requesting juice, they will be asked if there is an unavailable alternate flavor that he/she would prefer

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Driver, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States